CLINICAL TRIAL: NCT01129817
Title: Efficacy of Classification Based 'Cognitive Functional Therapy' in Patients With Non Specific Chronic Low Back Pain (NSCLBP) - A Randomized Controlled Trial
Brief Title: Efficacy of Classification Based 'Cognitive Functional Therapy' in Patients With Non Specific Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Kjartan Vibe Fersum, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 250.05.
Record Dates: First submitted 2010-05-20; First posted 2010-05-25 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Chronic Low Back Pain
Keywords: Cognitive Functional Therapy; Manual Therapy and Exercise; Chronic Low Back Pain; Randomized Controlled Trial; Subclassification
MeSH Terms: conditions — Motor Activity | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Functional Therapy (Experimental)
  Interventions: Other: Cognitive Functional Therapy
- Manual Therapy and Exercise (Active Comparator)
  Interventions: Other: Manual therapy and exercise

INTERVENTIONS:
Other: Cognitive Functional Therapy — A novel multidimensional classification system has been developed incorporating the biopsychosocial model, which subgroups patients based on their presentation with matched interventions directed at the maladaptive cognitive, physical and lifestyle behaviours associated with the disorder. The intervention is called 'cognitive functional therapy' as it directly challenges these behaviours in a functionally specific and graduated manner.
  Arms: Cognitive Functional Therapy
Other: Manual therapy and exercise — Patients in this group was treated with joint mobilization or manipulation techniques applied to the spine or pelvis primarily and was designed to be consistent with best current manual therapy practice in Norway. The particular dose and techniques were at the discretion of the treating therapist, based on each participant's objective and physical examination findings. In addition most of the patients in this group was given exercises or a home exercise program.
  Arms: Manual Therapy and Exercise

SUMMARY:
A randomized controlled trial of the efficacy of classification based cognitive functional physiotherapy according to the system proposed by Peter O'Sullivan as compared to manual therapy and exercise in patients with non specific chronic low back pain.

The investigators hypothesis was that treatment targeted at the mechanism behind the problem from a multidimensional perspective would be superior to traditional treatment.

DETAILED DESCRIPTION:
NSCLBP is widely viewed as a multifactorial biopsychosocial pain syndrome. It has been proposed by several authors that NSCLBP represents a vicious cycle associated with different combinations of maladaptive; cognitive (negative beliefs, fear avoidance behaviours, catastrophising, depression, stress, lack of pacing and coping), physical (pain provocative postures, movement patterns and pain behaviours) and lifestyle (inactivity, rest) behaviours that act to promote pain and disability. However a recent systematic review suggests that this change in paradigm and our new understanding of NSCLBP has not resulted in clinical trials utilizing multidimensional classification systems or targeted interventions based on the underlying mechanisms. line with this shift in paradigm a novel multidimensional classification system has been developed incorporating the biopsychosocial model, which subgroups patients based on their presentation of. with matched interventions directed at the maladaptive cognitive, physical and lifestyle behaviours associated with the disorder.

ELIGIBILITY:
Inclusion Criteria:

* all patients with non-specific LBP for more that 8 weeks duration
* mechanical provocation of pain with postures, movement and activities
* localised pain in the area from T12 to gluteal folds
* moderate ongoing LBP with a VAS > 2/10
* disability had to be higher than 14% on Oswestry Disability Index

Exclusion Criteria:

* sick listed for more than 4 months continuous duration
* acute exacerbation of LBP
* radicular pain with positive neural tissue provocation test
* any low limb surgery on the last 3 months
* surgery involving the lumbar spine (fusion)
* pregnancy
* psychiatric disorders - somatisation
* dominant psycho-social problems
* widespread non-specific pain disorder (no primary LBP focus)
* specific diagnoses: active rheumatologic disease, progressive neurological disease, serious cardiac or other internal medical condition, malignant basic diseases, acute traumas, infections, or acute vascular catastrophies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2006-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Pain | 12 months
  Pain was assessed using a pain numerical rating scale from 0 to 10
Disability | 12 months
  Disability measured by Oswestry Disability Index.

SECONDARY OUTCOMES:
Well being | 12 months
  Hopkins Symptoms Checklist.
Beliefs | 12 months
  Fear Avoidance Beliefs Questionnaire
Screening questionnaire | 12 months
  The Ørebro Pain Screening Questionnaire
Patient satisfaction | 12 months
  patient satisfaction. 5 items scale

CONTACTS AND LOCATIONS:
Overall Officials: Kjartan Vibe Fersum, PhD Student, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway

REFERENCES:
- [Derived] Vibe Fersum K, Smith A, Kvale A, Skouen JS, O'Sullivan P. Cognitive functional therapy in patients with non-specific chronic low back pain-a randomized controlled trial 3-year follow-up. Eur J Pain. 2019 Sep;23(8):1416-1424. doi: 10.1002/ejp.1399. Epub 2019 May 14. PMID 30974479